CLINICAL TRIAL: NCT02803580
Title: IPF Italian Observational Study (FIBRONET)
Brief Title: IPF Italian Observational Study (FIBRONET) in Idiopathic Pulmonary Fibrosis
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1199.262
Record Dates: First submitted 2015-11-30; First posted 2016-06-17 (Estimated); Results first posted 2019-09-13 (Actual); Last update posted 2019-09-13 (Actual); Status verified 2019-08

CONDITIONS: Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
The purpose of the present study is to evaluate the characteristics, management and clinical course of patients with IPF as treated under real-world in Italian Pulmonary Centres, in terms of symptoms, lung function and exercise tolerance during 12 months of observation.

ELIGIBILITY:
Inclusion criteria:

1. Patients aged>=40 years
2. Written informed consent to both participation in the study and privacy
3. Physician diagnosed IPF during the last 3 months based upon recent American Thoracic Society/European Resp. Society/Japanese Resp. Society/Latin American Thoracic Association guidelines 2011 (see Tables A1-A2 for High Resolution Chest Computer Tomography and histology criteria):

   * Exclusion of other known causes of Interstitial Lung Disease (e.g. domestic and occupational environmental exposures, connective tissue disease and drug toxicity)
   * Assessment of Idiopathic Pulmonary Fibrosis based on High Resolution Computed Tomography (HRCT) or HRCT and surgical lung biopsy if available.
4. Patient with further follow-up possible with enrolling investigator during planned study period
5. Patients capable of discernment and able to read or write in Italian language.

Exclusion criteria:

1. Inclusion in clinical trials or other IPF/ILD registries
2. Lung transplantation expected within the next 6 months
3. Pregnancy or breast feeding

Ages: 40 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: IPF pts
Sampling Method: Probability Sample
Enrollment: 209 (Actual)
Dates: Start 2015-11-17 (Actual); Primary Completion 2018-05-15 (Actual); Study Completion 2018-05-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (18):
- Italy (18):
  - A.O.U. Policlinico Vittorio Emanuele, Catania
  - Osp. Clin. SS. Anunziata, Chieti
  - Ospedale Colonnello D Avanzo, Foggia
  - Ospedale "G.B. Morgagni - L. Pierantoni" ausl forli, Forlì
  - Osp. S. Giuseppe Fatebenefratelli, Milan
  - Azienda Ospedaliera Policlinico di Modena, Modena
  - A.O. San Gerardo di Monza, Monza
  - Azienda Ospedaliera Universitaria "Federico II", Napoli
  - Azienda Sanitaria Ospedale S. Luigi Gonzaga, Orbassano
  - Azienda Ospedaliera Universitaria di Padova, Padua
  - Fondazione IRCCS Policlinico S. Matteo, Pavia
  - Ospedale di Cisanello, Pisa
  - Pol. Universitario Tor Vergata, Roma
  - A.O. San Camillo Forlanini, Roma
  - Policlinico Gemelli, Roma
  - Policlinico Universitario di Sassari, Sassari
  - A.O.U. Senese Policlinico Santa Maria alle Scotte, Siena
  - Ospedale Riuniti di Ancona, Torrette-Ancona

REFERENCES:
- [Derived] Poletti V, Vancheri C, Albera C, Harari S, Pesci A, Metella RR, Campolo B, Crespi G, Rizzoli S; FIBRONET study group. Clinical course of IPF in Italian patients during 12 months of observation: results from the FIBRONET observational study. Respir Res. 2021 Feb 24;22(1):66. doi: 10.1186/s12931-021-01643-w. PMID 33627105

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was an observational study based on participants newly diagnosed with Idiopathic Pulmonary Fibrosis (IPF) for less than 3 months, who enrolled in 20 Italian Pulmonary Centers highly experienced in the disease management of IPF. Data collection was performed between 30th November 2015 and 15th May 2018.
Pre-assignment Details: Data source for this study were medical records usually collected during routine clinical practice other than study-specific questionnaires.
Groups:
- Participants With Idiopathic Pulmonary Fibrosis: Participants with Idiopathic Pulmonary Fibrosis (IPF) as treated under real-world in Italian Pulmonary Centers, were enrolled between 30th November 2015 to 6th April 2017, followed by an observational phase of 12 months.
Period: Overall Study
Arm/Group | Participants With Idiopathic Pulmonary Fibrosis
Started | 209
Completed | 173
Not Completed | 36
Not completed — Death | 13
Not completed — Lost to Follow-up | 19
Not completed — Withdrawal by Subject | 3
Not completed — Inclusion in clinical trial | 1

BASELINE CHARACTERISTICS:
Population: All patients who enrolled in the Italian Pulmonary Centers from 30th November 2015 to 6th April 2017 were included.
Arm/Group | Participants With Idiopathic Pulmonary Fibrosis
Number analyzed (Participants) | 209
Age, Continuous [Mean (Standard Deviation); unit: Years] | 69.54 (7.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36
  Male | 173
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Ethnicity data were not collected from any participant.
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 209
  More than one race | 0
  Unknown or Not Reported | 0
IPF symptoms [Number; unit: Percentage of participants]
  More than 1 IPF symptom | 88.0
  Cough | 59.8
  Fatigue | 54.1
  Dizziness | 1.4
  Chest pain | 4.8
  Other | 20.1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With IPF Symptoms
Description: Percentage of participants with IPF symptoms such as cough, fatigue, dizziness, chest pain or any other symptom at 12-month follow up visit. The symptoms in the class 'other' reported upon specific visits were dyspnea, hemoptysis, post-nasal drip, sputum, weight loss, worsening of fatigue and lack of appetite.
  Baseline (V1), 3 months (V2), 6 months (V3), 9 months (V4) and 12 months (V5).
Time Frame: Baseline, 3 months, 6 months, 9 months and 12 months
Population: All participants who enrolled in the Italian Pulmonary Centers from 30th November 2015 to 6th April 2017 were included. Participants with values available at baseline and at follow up visits were considered.
Measure: Number; unit: Percentage of participants
Arm/Group | Participants With Idiopathic Pulmonary Fibrosis
Number analyzed (Participants) | 209
Percentage of participants
  More than 1 IPF symptom - V1 | 88.0
  More than 1 IPF symptom - V2: number analyzed (Participants) | 191
  More than 1 IPF symptom - V2 | 51.8
  More than 1 IPF symptom - V3: number analyzed (Participants) | 172
  More than 1 IPF symptom - V3 | 49.4
  More than 1 IPF symptom - V4: number analyzed (Participants) | 161
  More than 1 IPF symptom - V4 | 42.9
  More than 1 IPF symptom - V5: number analyzed (Participants) | 174
  More than 1 IPF symptom - V5 | 45.4
  Cough - V1 | 59.8
  Cough - V2: number analyzed (Participants) | 191
  Cough - V2 | 38.7
  Cough - V3: number analyzed (Participants) | 172
  Cough - V3 | 36.6
  Cough - V4: number analyzed (Participants) | 161
  Cough - V4 | 29.2
  Cough - V5: number analyzed (Participants) | 174
  Cough - V5 | 30.5
  Fatigue - V1 | 54.1
  Fatigue - V2: number analyzed (Participants) | 191
  Fatigue - V2 | 35.1
  Fatigue - V3: number analyzed (Participants) | 172
  Fatigue - V3 | 33.1
  Fatigue - V4: number analyzed (Participants) | 161
  Fatigue - V4 | 26.1
  Fatigue - V5: number analyzed (Participants) | 174
  Fatigue - V5 | 32.2
  Dizziness - V1 | 1.4
  Dizziness - V2: number analyzed (Participants) | 191
  Dizziness - V2 | 3.7
  Dizziness - V3: number analyzed (Participants) | 172
  Dizziness - V3 | 1.7
  Dizziness - V4: number analyzed (Participants) | 161
  Dizziness - V4 | 1.9
  Dizziness - V5: number analyzed (Participants) | 174
  Dizziness - V5 | 2.3
  Chest pain - V1 | 4.8
  Chest pain - V2: number analyzed (Participants) | 191
  Chest pain - V2 | 2.6
  Chest pain - V3: number analyzed (Participants) | 172
  Chest pain - V3 | 4.1
  Chest pain - V4: number analyzed (Participants) | 161
  Chest pain - V4 | 1.9
  Chest pain - V5: number analyzed (Participants) | 174
  Chest pain - V5 | 4.0
  Other - V1 | 20.1
  Other - V2: number analyzed (Participants) | 191
  Other - V2 | 8.4
  Other - V3: number analyzed (Participants) | 172
  Other - V3 | 5.2
  Other - V4: number analyzed (Participants) | 161
  Other - V4 | 6.2
  Other - V5: number analyzed (Participants) | 174
  Other - V5 | 5.2

2. Primary Outcome: Change From Baseline to Follow-up Visits in Lung Function: Vital Capacity
Description: In calculating the change from baseline to all follow-up visits (3 months, 6 months, 9 months and 12 months) in lung function: Vital Capacity (VC), only participants with values available at baseline and at follow up were considered. At follow up visit the absolute changes of lung function assessment vs baseline value was calculated as:
  Change in parameter VC = value of parameter VC at follow up visit - value of parameter VC at baseline visit.
  A positive value of change indicates a better outcome.
Time Frame: Baseline, 3 months, 6 months, 9 months and 12 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Liters (L)
Arm/Group | Participants With Idiopathic Pulmonary Fibrosis
Number analyzed (Participants) | 209
Liters (L)
  V2-V1: number analyzed (Participants) | 76
  V2-V1 | 0.08 (0.47)
  V3-V1: number analyzed (Participants) | 65
  V3-V1 | 0.07 (0.55)
  V4-V1: number analyzed (Participants) | 57
  V4-V1 | 0.07 (0.58)
  V5-V1: number analyzed (Participants) | 66
  V5-V1 | 0.03 (0.58)

3. Primary Outcome: Change From Baseline to Follow-up Visits in Lung Function: Forced Vital Capacity (Actual)
Description: In calculating the change from baseline to follow-up visits in lung function: Forced Vital Capacity (FVC), only participants with values available at baseline and at follow up were considered. At follow up visit the absolute changes of lung function assessment vs baseline value was calculated as:
  Change in parameter FVC = value of parameter FVC at follow up visit - value of parameter FVC at baseline visit.
  A positive value of change indicates a better outcome.
Time Frame: Baseline, 3 months, 6 months, 9 months and 12 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Participants With Idiopathic Pulmonary Fibrosis
Number analyzed (Participants) | 209
L
  V2-V1 Actual: number analyzed (Participants) | 159
  V2-V1 Actual | -0.02 (0.27)
  V3-V1 Actual: number analyzed (Participants) | 144
  V3-V1 Actual | -0.02 (0.34)
  V4-V1 Actual: number analyzed (Participants) | 120
  V4-V1 Actual | -0.02 (0.31)
  V5-V1 Actual: number analyzed (Participants) | 136
  V5-V1 Actual | -0.05 (0.33)

4. Primary Outcome: Change From Baseline to Follow-up Visits in Lung Function: Forced Vital Capacity (Predicted)
Description: In calculating the change from baseline to follow-up visits in lung function: Forced Vital Capacity (FVC), only participants with values available at baseline and at follow up were considered. At follow up visit the absolute changes of lung function assessment vs baseline value was calculated as:
  Change in parameter FVC = value of parameter FVC at follow up visit - value of parameter FVC at baseline visit.
  A positive value of change indicates a better outcome.
  The value of FVC % of predicted is a relevant parameter to understand and classify the severity of the disease at the diagnosis and to follow up patients during the treatment (i.e. annual rate decline of FVC >10% is a predictor of high rate of mortality).
Time Frame: Baseline, 3 months, 6 months, 9 months and 12 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent Predicted
Arm/Group | Participants With Idiopathic Pulmonary Fibrosis
Number analyzed (Participants) | 209
Percent Predicted
  V2-V1 Predicted | 0.31 (8.82)
  V3-V1 Predicted | 1.59 (8.20)
  V4-V1 Predicted | 1.36 (9.39)
  V5-V1 Predicted | 0.01 (10.17)

5. Primary Outcome: Change From Baseline to Follow-up Visits in Lung Function: Forced Expiratory Volume in the 1st Second
Description: In calculating the change from baseline to follow-up visits in lung function: Forced Expiratory Volume in the 1st second (FEV1), only participants with values available at baseline and at follow up were considered. At follow up visit the absolute changes of lung function assessment vs baseline value was calculated as:
  Change in parameter FEV1 = value of parameter FEV1 at follow up visit - value of parameter FEV1 at baseline visit.
  A positive value of change indicates a better outcome.
Time Frame: Baseline, 3 months, 6 months, 9 months and 12 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Participants With Idiopathic Pulmonary Fibrosis
Number analyzed (Participants) | 209
L
  V2-V1: number analyzed (Participants) | 159
  V2-V1 | 0.01 (0.21)
  V3-V1: number analyzed (Participants) | 143
  V3-V1 | -0.02 (0.22)
  V4-V1: number analyzed (Participants) | 120
  V4-V1 | -0.01 (0.24)
  V5-V1: number analyzed (Participants) | 135
  V5-V1 | -0.02 (0.28)

6. Primary Outcome: Change From Baseline to Follow-up Visits in Lung Function: Total Lung Capacity
Description: In calculating the change from baseline to follow-up visits in lung function: Total Lung Capacity (TLC), only participants with values available at baseline and at follow up were considered. At follow up visit the absolute changes of lung function assessment vs baseline value was calculated as:
  Change in parameter TLC = value of parameter TLC at follow up visit - value of parameter TLC at baseline visit.
  A positive value of change indicates a better outcome.
Time Frame: Baseline, 3 months, 6 months, 9 months and 12 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Participants With Idiopathic Pulmonary Fibrosis
Number analyzed (Participants) | 209
L
  V2-V1: number analyzed (Participants) | 96
  V2-V1 | -0.07 (0.62)
  V3-V1: number analyzed (Participants) | 97
  V3-V1 | -0.05 (0.72)
  V4-V1: number analyzed (Participants) | 72
  V4-V1 | -0.03 (0.65)
  V5-V1: number analyzed (Participants) | 89
  V5-V1 | -0.11 (0.65)

7. Primary Outcome: Change From Baseline to Follow-up Visits in Lung Function: Diffusion Capacity for Carbon Monoxide
Description: In calculating the change from baseline to follow-up visits in lung function: Diffusion capacity for carbon monoxide (DLCO), only participants with values available at baseline and at follow up were considered. At follow up visit the absolute changes of lung function assessment vs baseline value was calculated as:
  Change in parameter DLCO = value of parameter DLCO at follow up visit - value of parameter DLCO at baseline visit.
  A positive value of change indicates a better outcome.
  Values of DLCO with unit = milliliter/minute/millimeter mercury (ml/min/mmHg) were converted to micromole/minute/kilopascal (mmol/min/kPa) according to the following formula:
  DLCO (mmol/min/kPa) = DLCO (ml/min/mmHg)/2.986 [46].
Time Frame: Baseline, 3 months, 6 months, 9 months and 12 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/min/kPa
Arm/Group | Participants With Idiopathic Pulmonary Fibrosis
Number analyzed (Participants) | 209
mmol/min/kPa
  V2-V1: number analyzed (Participants) | 121
  V2-V1 | -0.41 (2.52)
  V3-V1: number analyzed (Participants) | 116
  V3-V1 | -0.46 (2.27)
  V4-V1: number analyzed (Participants) | 92
  V4-V1 | -0.34 (2.97)
  V5-V1: number analyzed (Participants) | 99
  V5-V1 | -0.25 (3.03)

8. Primary Outcome: Change From Baseline to Follow-up Visits in Lung Function: Partial Pressure of Oxygen
Description: In calculating the change from baseline to follow-up visits in lung function: Partial Pressure of Oxygen (PO2), only participants with values available at baseline and at follow up were considered. At follow up visit the absolute changes of lung function assessment vs baseline value was calculated as:
  Change in parameter PO2 = value of parameter PO2 at follow up visit - value of parameter PO2 at baseline visit.
  A positive value of change indicates a better outcome.
Time Frame: Baseline, 3 months, 6 months, 9 months and 12 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Millimeter mercury (mmHg)
Arm/Group | Participants With Idiopathic Pulmonary Fibrosis
Number analyzed (Participants) | 209
Millimeter mercury (mmHg)
  V2-V1: number analyzed (Participants) | 31
  V2-V1 | -0.06 (6.22)
  V3-V1: number analyzed (Participants) | 29
  V3-V1 | 2.13 (9.56)
  V4-V1: number analyzed (Participants) | 18
  V4-V1 | 1.11 (9.88)
  V5-V1: number analyzed (Participants) | 29
  V5-V1 | -0.47 (14.05)

9. Primary Outcome: Change From Baseline to Follow-up Visits in Lung Function: Partial Pressure of Carbon Dioxide
Description: In calculating the change from baseline to follow-up visits in lung function: Partial Pressure of Carbon dioxide (PCO2), only patients with values available at baseline and at follow up were considered. At follow up visit the absolute changes of lung function assessment vs baseline value was calculated as:
  Change in parameter PCO2 = value of parameter PCO2 at follow up visit - value of parameter PCO2 at baseline visit.
  A positive value of change indicates a better outcome.
Time Frame: Baseline, 3 months, 6 months, 9 months and 12 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Participants With Idiopathic Pulmonary Fibrosis
Number analyzed (Participants) | 209
mmHg
  V2-V1: number analyzed (Participants) | 30
  V2-V1 | 1.03 (3.63)
  V3-V1: number analyzed (Participants) | 29
  V3-V1 | 1.59 (5.36)
  V4-V1: number analyzed (Participants) | 18
  V4-V1 | 1.24 (4.42)
  V5-V1: number analyzed (Participants) | 29
  V5-V1 | 1.12 (3.75)

10. Primary Outcome: Change From Baseline to Follow-up Visits in Lung Function: Oxygen Saturation
Description: In calculating the change from baseline to follow-up visits in lung function: Oxygen Saturation (SaO2), only participants with values available at baseline and at follow up were considered. At follow up visit the absolute changes of lung function assessment vs baseline value was calculated as:
  Change in parameter SaO2 = value of parameter SaO2 at follow up visit - value of parameter SaO2 at baseline visit.
  A positive value of change indicates a better outcome.
Time Frame: Baseline, 3 months, 6 months, 9 months and 12 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage (%) of SaO2
Arm/Group | Participants With Idiopathic Pulmonary Fibrosis
Number analyzed (Participants) | 209
Percentage (%) of SaO2
  V2-V1: number analyzed (Participants) | 128
  V2-V1 | -0.05 (2.05)
  V3-V1: number analyzed (Participants) | 121
  V3-V1 | -0.33 (2.23)
  V4-V1: number analyzed (Participants) | 97
  V4-V1 | -0.02 (2.27)
  V5-V1: number analyzed (Participants) | 107
  V5-V1 | -0.13 (2.56)

11. Primary Outcome: Change From Baseline to Follow-up Visits in Lung Function: Partial Pressure of Oxygen in Arterial Blood at Rest
Description: In calculating the change from baseline to follow-up visits in lung function: Partial Pressure of Oxygen in arterial blood at rest (PaO2), only participants with values available at baseline and at follow up were considered. At follow up visit the absolute changes of lung function assessment vs baseline value was calculated as:
  Change in parameter PaO2 = value of parameter PaO2 at follow up visit - value of parameter PaO2 at baseline visit.
  A positive value of change indicates a better outcome.
Time Frame: Baseline, 3 months, 6 months, 9 months and 12 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Participants With Idiopathic Pulmonary Fibrosis
Number analyzed (Participants) | 209
mmHg
  V2-V1: number analyzed (Participants) | 12
  V2-V1 | -0.03 (6.78)
  V3-V1: number analyzed (Participants) | 12
  V3-V1 | 2.74 (5.44)
  V4-V1: number analyzed (Participants) | 11
  V4-V1 | -0.60 (4.48)
  V5-V1: number analyzed (Participants) | 9
  V5-V1 | 1.43 (4.86)

12. Primary Outcome: Change From Baseline to Follow-up Visits in Lung Function: Partial Pressure of Carbon Dioxide in Arterial Blood at Rest
Description: In calculating the change from baseline to follow-up visits in lung function: Partial Pressure of Carbon dioxide in arterial blood at rest (PaCO2), only participants with values available at baseline and at follow up were considered. At follow up visit the absolute changes of lung function assessment vs baseline value was calculated as:
  Change in parameter PaCO2 = value of parameter PaCO2 at follow up visit - value of parameter PaCO2 at baseline visit.
  A positive value of change indicates a better outcome.
Time Frame: Baseline, 3 months, 6 months, 9 months and 12 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Participants With Idiopathic Pulmonary Fibrosis
Number analyzed (Participants) | 209
mmHg
  V2-V1: number analyzed (Participants) | 12
  V2-V1 | 1.12 (2.98)
  V3-V1: number analyzed (Participants) | 12
  V3-V1 | 1.61 (2.63)
  V4-V1: number analyzed (Participants) | 11
  V4-V1 | 0.65 (2.99)
  V5-V1: number analyzed (Participants) | 9
  V5-V1 | 1.27 (4.20)

13. Primary Outcome: Change From Baseline to Follow-up Visits in Exercise Tolerance
Description: Change from baseline to follow-up visits in exercise tolerance was evaluated by means of change in 6 minute walked distance test.
  Change versus baseline was calculated as parameter at follow up - parameter at baseline.
  A positive value of change indicates a better outcome. The 6-minute walked distance test was carried out using two parameters start of peripheral capillary oxygen saturation (SpO2) and SpO2 at the end of the test. Only participants with values available at baseline and at follow up were considered
Time Frame: Baseline, 3 months, 6 months, 9 months and 12 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage (%) of SpO2
Arm/Group | Participants With Idiopathic Pulmonary Fibrosis
Number analyzed (Participants) | 209
Percentage (%) of SpO2
  SpO2 at start of the test - V2-V1: number analyzed (Participants) | 77
  SpO2 at start of the test - V2-V1 | 0.11 (1.99)
  SpO2 at start of the test - V3-V1: number analyzed (Participants) | 77
  SpO2 at start of the test - V3-V1 | 0.11 (1.96)
  SpO2 at start of the test - V4-V1: number analyzed (Participants) | 71
  SpO2 at start of the test - V4-V1 | -0.04 (2.03)
  SpO2 at start of the test - V5-V1: number analyzed (Participants) | 75
  SpO2 at start of the test - V5-V1 | 0.16 (1.69)
  SpO2 at the end of the test - V2-V1: number analyzed (Participants) | 77
  SpO2 at the end of the test - V2-V1 | -0.52 (3.23)
  SpO2 at the end of the test - V3-V1: number analyzed (Participants) | 77
  SpO2 at the end of the test - V3-V1 | -0.64 (2.88)
  SpO2 at the end of the test - V4-V1: number analyzed (Participants) | 71
  SpO2 at the end of the test - V4-V1 | 0.07 (5.32)
  SpO2 at the end of the test - V5-V1: number analyzed (Participants) | 75
  SpO2 at the end of the test - V5-V1 | 0.19 (3.21)

14. Secondary Outcome: Characteristic of Participants at Enrollment: Key Socio-demographic Data: Age
Description: IPF enrolled participants were described in terms of socio-demographic variables (e.g. age, gender, race, body mass index, educational degree, and employment status) at baseline.
Time Frame: Baseline
Population: All participants who enrolled in the Italian Pulmonary Centers from 30th November 2015 to 6th April 2017 were included.
Measure: Mean (Standard Deviation); unit: Years
Arm/Group | Participants With Idiopathic Pulmonary Fibrosis
Number analyzed (Participants) | 209
Years | 69.54 (7.43)

15. Secondary Outcome: Characteristic of Participants at Enrollment: Key Demographic Data: Gender
Description: IPF enrolled participants were described in terms of socio-economic variables; number of participants as per their gender are presented. The data is provided in baseline section.
Time Frame: Baseline
Population: All participants who enrolled in the Italian Pulmonary Centers from 30th November 2015 to 6th April 2017 were included.
Measure: Number; unit: Participants
Arm/Group | Participants With Idiopathic Pulmonary Fibrosis
Number analyzed (Participants) | 209
Participants
  Male | 173
  Female | 36

16. Secondary Outcome: Characteristic of Participants at Enrollment: Key Demographic Data: Race
Description: IPF enrolled participants were described in terms of socio-economic variables; number of participants as per their race are presented. The data is provided in baseline section.
Time Frame: Baseline
Population: All participants who enrolled in the Italian Pulmonary Centers from 30th November 2015 to 6th April 2017 were included.
Measure: Number; unit: Participants
Arm/Group | Participants With Idiopathic Pulmonary Fibrosis
Number analyzed (Participants) | 209
Participants
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 209
  More than one race | 0
  Unknown or Not Reported | 0

17. Secondary Outcome: Characteristic of Participants at Enrollment: Key Demographic Data: Highest Education Level
Description: IPF enrolled participants were described in terms of socio-economic variables; number of participants as per their highest education level.
Time Frame: Baseline
Population: All participants who enrolled in the Italian Pulmonary Centers from 30th November 2015 to 6th April 2017 were included.
Measure: Number; unit: Participants
Arm/Group | Participants With Idiopathic Pulmonary Fibrosis
Number analyzed (Participants) | 209
Participants
  None | 1
  Primary School | 34
  Middle school | 55
  High school | 45
  Academic degree | 20
  Unknown | 54

18. Secondary Outcome: Characteristic of Participants at Enrollment: Key Demographic Data: Employment Status
Description: IPF enrolled participants were described in terms of socio-economic variables; number of participants as per their employment status are presented.
Time Frame: Baseline
Population: All participants who enrolled in the Italian Pulmonary Centers from 30th November 2015 to 6th April 2017 were included.
Measure: Number; unit: Participants
Arm/Group | Participants With Idiopathic Pulmonary Fibrosis
Number analyzed (Participants) | 209
Participants
  Unemployed | 9
  Employed | 51
  Retired | 130
  Housewife / househusband | 14
  Unknown | 5

19. Secondary Outcome: Characteristic of IPF Patients at Enrollment: Key Demographic Data: Body Mass Index
Description: IPF enrolled participants were described in terms of socio-economic variables; number of participants as per their Body mass index are presented.
Time Frame: Baseline
Population: All participants who enrolled in the Italian Pulmonary Centers from 30th November 2015 to 6th April 2017 were included.
Measure: Number; unit: Participants
Arm/Group | Participants With Idiopathic Pulmonary Fibrosis
Number analyzed (Participants) | 209
Participants
  Underweight | 2
  Normal weight | 34
  Overweight | 81
  Obese | 50
  Not Reported | 42

20. Secondary Outcome: Characteristic of Participants at Enrollment: Key Demographic Data: Housing Situation
Description: IPF enrolled participants were described in terms of socio-economic variables; number of participants as per their housing situation are presented.
Time Frame: Baseline
Population: All participants who enrolled in the Italian Pulmonary Centers from 30th November 2015 to 6th April 2017 were included.
Measure: Number; unit: Participants
Arm/Group | Participants With Idiopathic Pulmonary Fibrosis
Number analyzed (Participants) | 209
Participants
  Home (alone) | 11
  Home (with family) | 182
  Institution | 2
  Unknown | 14

21. Secondary Outcome: Characteristic of Participants at Enrollment: Key Demographic Data: Marital Status
Description: IPF enrolled participants were described in terms of socio-economic variables; number of participants as per their marital status are presented.
Time Frame: Baseline
Population: All participants who enrolled in the Italian Pulmonary Centers from 30th November 2015 to 6th April 2017 were included.
Measure: Number; unit: Participants
Arm/Group | Participants With Idiopathic Pulmonary Fibrosis
Number analyzed (Participants) | 209
Participants
  Married | 169
  Single | 9
  Widow / Widowed | 9
  Unknown | 22

22. Secondary Outcome: IPF Risk Factors: Smoking Habit
Description: IPF enrolled participants were described in terms of potential IPF risk factors; number of participants as per their smoking habits are presented.
Time Frame: Baseline
Population: All participants who enrolled in the Italian Pulmonary Centers from 30th November 2015 to 6th April 2017 were included.
Measure: Number; unit: Participants
Arm/Group | Participants With Idiopathic Pulmonary Fibrosis
Number analyzed (Participants) | 209
Participants
  Former smokers | 138
  Current smokers | 9
  No smokers | 62

23. Secondary Outcome: IPF Risk Factors: Environmental Exposure
Description: IPF enrolled participants were described in terms of potential IPF risk factors; number of participants as per their environmental exposure (such as bricklayer, building material dust, cement dust, chemical gas, coal dust, factory food, marble dust, masonry dust, mold, paint, powdered detergent and textile material) are presented.
Time Frame: Baseline
Population: All participants who enrolled in the Italian Pulmonary Centers from 30th November 2015 to 6th April 2017 were included.
Measure: Number; unit: Participants
Arm/Group | Participants With Idiopathic Pulmonary Fibrosis
Number analyzed (Participants) | 209
Participants
  No | 136
  Yes | 70
  Unknown | 3

24. Secondary Outcome: IPF Risk Factors: Exposure to Drugs Associated With IPF
Description: IPF enrolled participants were described in terms of potential IPF risk factors; number of participants as per their exposure to drugs associated with IPF are presented.
Time Frame: Baseline
Population: All participants who enrolled in the Italian Pulmonary Centers from 30th November 2015 to 6th April 2017 were included.
Measure: Number; unit: Participants
Arm/Group | Participants With Idiopathic Pulmonary Fibrosis
Number analyzed (Participants) | 209
Participants
  Drug Exposure - Amiodarone | 2
  No drug exposure | 207

25. Secondary Outcome: IPF Risk Factors: Family History
Description: IPF enrolled participants were described in terms of potential IPF risk factors; number of participants as per their family history for IPF are presented.
Time Frame: Baseline
Population: All participants who enrolled in the Italian Pulmonary Centers from 30th November 2015 to 6th April 2017 were included.
Measure: Number; unit: Participants
Arm/Group | Participants With Idiopathic Pulmonary Fibrosis
Number analyzed (Participants) | 209
Participants
  No | 183
  Yes | 25
  Unknown | 1

26. Secondary Outcome: Number of Participants With Comorbidity
Description: Number of participants with ongoing comorbidities (such as gastroesophageal reflux disease, pulmonary hypertension, emphysema, lung cancer, coronary heart disease, depression) are provided. Some participants reported more than one comorbidity at enrollment.
Time Frame: Baseline
Population: All participants who enrolled in the Italian Pulmonary Centers from 30th November 2015 to 6th April 2017 were included.
Measure: Number; unit: Participants
Arm/Group | Participants With Idiopathic Pulmonary Fibrosis
Number analyzed (Participants) | 209
Participants
  Anxiety/Depression | 12
  Arterial hypertension | 103
  Atherothrombotic disease | 27
  Atrial fibrillation | 9
  Benign Prostatic Hypertrophy | 25
  Cerebrovascular disease (Carotid stenosis, stroke) | 13
  Deep venous thrombosis | 1
  Diabetes mellitus | 45
  Emphysema | 8
  Gastroesophageal reflux disease | 49
  Hypercholesterolemia | 17
  Lung cancer | 1
  Peripheral arterial disease | 2
  Pulmonary hypertension | 6
  Renal insufficiency | 5
  Other | 80
  Previous myocardial infarction | 23

27. Secondary Outcome: IPF Disease Severity and Manifestation
Description: IPF disease severity and manifestation (including lung function, cardiopulmonary exercise testing and/or exercise capacity if available, laboratory values) is measured by the FVC. Percentages are calculated out of the total number of evaluable participants with available FVC of the predicted at baseline.
Time Frame: Baseline
Population: All participants who enrolled in the Italian Pulmonary Centers from 30th November 2015 to 6th April 2017 were included.
Measure: Number; unit: Percentage of participants
Arm/Group | Participants With Idiopathic Pulmonary Fibrosis
Number analyzed (Participants) | 196
Percentage of participants
  FVC <50% | 4.1
  FVC between 50%-70% | 24.5
  FVC between 70%-90% | 41.3
  FVC >=90% | 30.1

28. Secondary Outcome: Number of Participants With Different Methods Used for IPF Diagnosis
Description: Several diagnostic approaches were used to detect IPF, the main ones being High Resolution chest Computer Tomography (HRCT), surgical lung biopsy, Bronchoalveolar lavage (BAL), transbronchial biopsy and spirometry.
Time Frame: Baseline
Population: All participants who enrolled in the Italian Pulmonary Centers from 30th November 2015 to 6th April 2017 were included.
Measure: Number; unit: Participants
Arm/Group | Participants With Idiopathic Pulmonary Fibrosis
Number analyzed (Participants) | 209
Participants
  HRCT | 209
  Surgical lung biopsy | 14
  BAL | 40
  Transbronchial Biopsy | 11
  Spirometry | 58
  Other | 27

29. Secondary Outcome: IPF Treatment Modalities: Non-pharmacological Treatment
Description: Number of participants with ≥1 non-pharmacological therapy for IPF ongoing at baseline (visit 1), 3-month (visit 2), 6-month (visit 3) and 12-month (visit 5) follow up visits are presented.
Time Frame: Baseline, 3 months, 6 months and 12 months
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Participants With Idiopathic Pulmonary Fibrosis
Number analyzed (Participants) | 209
Participants
  V1: Long-term oxygen therapy (LtOT) | 7
  V2: LtOT-Cardiopulmonary exercise training: number analyzed (Participants) | 191
  V2: LtOT-Cardiopulmonary exercise training | 1
  V2: LtOT: number analyzed (Participants) | 191
  V2: LtOT | 15
  V3: LtOT: number analyzed (Participants) | 172
  V3: LtOT | 12
  V3: LtOT-Cardiopulmonary exercise training: number analyzed (Participants) | 172
  V3: LtOT-Cardiopulmonary exercise training | 2
  V5: LtOT: number analyzed (Participants) | 174
  V5: LtOT | 13
  V5: LtOT-Cardiopulmonary exercise training: number analyzed (Participants) | 174
  V5: LtOT-Cardiopulmonary exercise training | 2

30. Secondary Outcome: IPF Treatment Modalities: Lung Transplantation
Description: Number of participants who had lung transplantation at baseline, 3-month, 6-month and 12-month follow up visits are presented.
Time Frame: Baseline, 3 months, 6 months and 12 months
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Participants With Idiopathic Pulmonary Fibrosis
Number analyzed (Participants) | 209
Participants
  V1 | 0
  V2: number analyzed (Participants) | 191
  V2 | 5
  V3: number analyzed (Participants) | 172
  V3 | 2
  V5: number analyzed (Participants) | 174
  V5 | 1

31. Secondary Outcome: IPF Treatment Modalities: Prescribed Drugs and Dose
Description: IPF Patients with ≥1 pharmacological therapy for IPF ongoing at baseline, 3-month, 6-month and 12-month follow up visits are presented. The pharmacological therapies used for IPF treatment are Nintedanib and Pirfenidone.
Time Frame: Baseline, 3 months, 6 months and 12 months
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Participants With Idiopathic Pulmonary Fibrosis
Number analyzed (Participants) | 209
Participants
  V1 | 33
  V2: number analyzed (Participants) | 191
  V2 | 138
  V3: number analyzed (Participants) | 172
  V3 | 139
  V5: number analyzed (Participants) | 174
  V5 | 146

32. Secondary Outcome: Number of Exacerbations During 12 Months of Observation
Description: Number of participants with mild, moderate and severe exacerbations during the observation period are presented. An exacerbation was considered occurred during observation period if onset date ≥ date of first IPF diagnosis and onset date ≤ last available visit date (for participants who completed the study) or date of drop out or date of death (for participants who did not complete the study).
Time Frame: Up to 12 months
Population: All participants who enrolled in the Italian Pulmonary Centers from 30th November 2015 to 6th April 2017 were included.
Measure: Number; unit: Participants
Arm/Group | Participants With Idiopathic Pulmonary Fibrosis
Number analyzed (Participants) | 209
Participants
  Mild exacerbation | 7
  Moderate exacerbation | 7
  Severe exacerbation | 4

33. Secondary Outcome: Health Related Quality of Life Variation Measured With Saint George's Respiratory Questionnaire
Description: Health Related Quality of Life (HRQoL) variation measured with Saint George's Respiratory Questionnaire (SGRQ), developed to measure health in chronic airflow limitation. It is a disease-specific instrument designed to measure health impairment in terms of impact on overall health, daily life, and perceived well-being in participants with obstructive airways disease. Three component scores (symptoms, activity and impacts on daily life) and a total score were calculated, with lower scores corresponding to better health. The Total score is calculated by summing all positive responses in the questionnaire and expressing the result as a percentage of overall impairment where 100 represents worst possible health status and 0 indicates best possible health status.
Time Frame: Baseline, 6 months and 12 months
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Unit on scale
Arm/Group | Participants With Idiopathic Pulmonary Fibrosis
Number analyzed (Participants) | 209
Unit on scale
  V1: number analyzed (Participants) | 181
  V1 | 39.82 [23.40 to 56.79]
  V3: number analyzed (Participants) | 137
  V3 | 41.14 [24.48 to 55.79]
  V5: number analyzed (Participants) | 134
  V5 | 39.60 [23.80 to 56.77]

34. Secondary Outcome: HRQoL Variation Measured With EuroQol Descriptive System
Description: The quality of life was evaluated by the EuroQol 5-dimension 5-level (EQ-5D-5L) a standardized measure of health status developed by EuroQol Group to provide a simple generic measure of health status for clinical and economic evaluation. EQ-5D-5L was filled in by participants, it was easy from a cognitive point of view, since it took only few minutes for filling. EQ-5D-5L consists of 2 sections: "EQ-5D descriptive system" and EQ visual analogue scale (EQ VAS). The EQ-5D-5L descriptive system comprises the following 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression.
Time Frame: Baseline, 6 months and 12 months
Population: as for outcome 1
Measure: Number; unit: Percentage (%) of participants
Arm/Group | Participants With Idiopathic Pulmonary Fibrosis
Number analyzed (Participants) | 209
Percentage (%) of participants
  Autonomous in self care - V1: number analyzed (Participants) | 205
  Autonomous in self care - V1 | 74.6
  Walk without difficulties - V1: number analyzed (Participants) | 205
  Walk without difficulties - V1 | 45.4
  Perform daily activies easily - V1: number analyzed (Participants) | 205
  Perform daily activies easily - V1 | 49.3
  Not to have pain - V1: number analyzed (Participants) | 205
  Not to have pain - V1 | 46.8
  Not to be anxious - V1: number analyzed (Participants) | 205
  Not to be anxious - V1 | 46.8
  Autonomous in self care - V3: number analyzed (Participants) | 160
  Autonomous in self care - V3 | 73.1
  Walk without difficulties - V3: number analyzed (Participants) | 160
  Walk without difficulties - V3 | 46.9
  Perform daily activies easily - V3: number analyzed (Participants) | 160
  Perform daily activies easily - V3 | 51.3
  Not to have pain - V3: number analyzed (Participants) | 160
  Not to have pain - V3 | 51.9
  Not to be anxious - V3: number analyzed (Participants) | 160
  Not to be anxious - V3 | 40.0
  Autonomous in self care - V5: number analyzed (Participants) | 157
  Autonomous in self care - V5 | 65.0
  Walk without difficulties - V5: number analyzed (Participants) | 157
  Walk without difficulties - V5 | 49.0
  Perform daily activies easily - V5: number analyzed (Participants) | 157
  Perform daily activies easily - V5 | 45.2
  Not to have pain - V5: number analyzed (Participants) | 157
  Not to have pain - V5 | 52.2
  Not to be anxious - V5: number analyzed (Participants) | 157
  Not to be anxious - V5 | 46.5

35. Secondary Outcome: HRQoL Measured With EQ VAS
Description: The quality of life was evaluated by the EQ-5D-5L a standardized measure of health status developed by EuroQol Group to provide a simple generic measure of health status for clinical and economic evaluation. EQ-5D-5L consists of 2 sections: "EQ-5D descriptive system" and EQ VAS. The EQ VAS indicate the health status self-assessed by the participants on a visual analogue scale from 0 to 100, where 100 is the "best imaginable health state" and 0 the "worst imaginable health state". It can be used as a quantitative measure of health as judged by participants.
Time Frame: Baseline, 6 months and 12 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Unit on scale
Arm/Group | Participants With Idiopathic Pulmonary Fibrosis
Number analyzed (Participants) | 157
Unit on scale
  V1 | 67.01 (18.29)
  V3 | 68.92 (16.12)
  V5 | 67.46 (17.75)

36. Secondary Outcome: Health Care Resource Consumption From Diagnosis up to End of 12 Months Follow-up According to the Italian National Health Service (INHS)
Description: The health care sector-related costs at diagnosis and from diagnosis up to the end of 12-month follow-up according to the INHS point of view, was carried out in a two-step approach:
  (i)First of all the resource consumption exclusively related to both IPF, IPF exacerbations and IPF-related adverse events since diagnosis was collected or estimated and then (ii) A monetary value was assigned to the collected or estimated resource consumption.
  Health care resource consumption was computed during observational period in terms of number of (inward and day-hospital) hospitalizations and number of Intensive Care Unit (ICU) admissions.
Time Frame: Up to 12 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Participants With Idiopathic Pulmonary Fibrosis
Number analyzed (Participants) | 209
Days
  Overall duration of inward hospitalization: number analyzed (Participants) | 13
  Overall duration of inward hospitalization | 14.92 (9.07)
  Overall duration of day-hospital hospitalization: number analyzed (Participants) | 0
  Overall duration of ICU admissions: number analyzed (Participants) | 1
  Overall duration of ICU admissions | 1 (NA) — Only one participant is involved.

ADVERSE EVENTS:
Time Frame: For serious adverse event (SAE) and Non-SAE: From IPF diagnosis until the end of observation period, up to 12 months. For All-cause mortality: From signing informed consent until the end of observation period, up to 493 days.
Description: All patients who enrolled in the Italian Pulmonary Centers from 30th November 2015 to 6th April 2017 were included.
Arm/Group | Participants With Idiopathic Pulmonary Fibrosis
All-Cause Mortality (participants affected / at risk) | 13/209
Serious Adverse Events (participants affected / at risk) | 16/209
Other Adverse Events (participants affected / at risk) | 38/209
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Participants With Idiopathic Pulmonary Fibrosis (N=209)
Angina pectoris (Cardiac disorders) | 1
Cardiac arrest (Cardiac disorders) | 3
Cardiac failure (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
Death (General disorders) | 3
Pneumonia (Infections and infestations) | 1
Epilepsy (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Participants With Idiopathic Pulmonary Fibrosis (N=209)
Diarrhoea (Gastrointestinal disorders) | 25
Rash (Skin and subcutaneous tissue disorders) | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-01-30): https://cdn.clinicaltrials.gov/large-docs/80/NCT02803580/SAP_000.pdf
  • Study Protocol (2015-06-26): https://cdn.clinicaltrials.gov/large-docs/80/NCT02803580/Prot_001.pdf